CLINICAL TRIAL: NCT03565692
Title: Lum-Iva-biota: Exploring the Respiratory Mycobiota and Microbiota Profile in French CF Patients Taking Lumacaftor-Ivacaftor
Acronym: Lum-Iva-Biota
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Societe Francaise de la Mucoviscidose (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2016/22
Record Dates: First submitted 2018-05-31; First posted 2018-06-21 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Cystic Fibrosis
Keywords: Microbiome; Microbiota; Mycobiota; Mycobiome; Deep-Sequencing; Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Human sputum and stool specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated by LUMACAFTOR-IVACAFTOR: Patients treated by LUMACAFTOR-IVACAFTOR (or other ivacaftor combinations) Patients over 6 years who are currently able to benefit from LUMACAFTOR-IVACAFTOR (or other ivacaftor combinations) according the mutation eligibility criteria and for whom conventional microbiological analysis of sputum samples and stool will be collected during their follow-up after the treatment onset.
  Interventions: Biological: the lung mycobiota and microbiota profile; Biological: the gut mycobiota and microbiota profile

INTERVENTIONS:
Biological: the lung mycobiota and microbiota profile — All sputum samples will follow regarding mycological and metagenomic analyses as summarized :
  * Pre-analytical treatment combining pre-treatment with mucolytic agent and sonication action
  * Separation of the pellet and supernatant, stored at -20 ° C until testing
  * Galactomannan (GM) Assay on each sputum supernatant to correlate with Aspergillus colonization history
  * Targeted metagenomics of bacterial communities (based on 16S amplification) and of fungal community (based on ITS2 amplification)
  * Bioinformatic analysis of metagenomics raw data, correlation with bioclinical data of each patient, statistical analysis, and characterization of phenomena of co-evolution/co-exclusion according to evolutionary ecology concepts.
  * Pseudomonas aeruginosa load measured by qPCR
Biological: the gut mycobiota and microbiota profile — All stool samples will follow regarding mycological and metagenomic analyses as summarized : - Separation of the pellet and supernatant, stored at -20 ° C until testing - Targeted metagenomics of bacterial communities (based on 16S amplification) and of fungal community (based on ITS2 amplification) - Bioinformatic analysis of metagenomics raw data, correlation with bioclinical data of each patient, statistical analysis, and characterization of phenomena of co-evolution/co-exclusion according to evolutionary ecology concepts. - Measurement of inflammation.

SUMMARY:
n2015, VERTEX company - producing already KALYDECO (IVACAFTOR, VX-770) potentiator molecule that is recommended for the treatment of CF patients aged ≥ 6 y, with CFTR mutation altering the channel regulation (class III mutations) as G551D, G1244E, G1349D, G178R, G551S, S1251N, S1255P, S549Nou S549R) -was allowed by the Federal Drug Administration (FDA) and European Medicines Agency (EMEA) for producing and using ivacaftor combination (such as lumacaftor/ ivacaftor initially, and more recently tezacaftor/ivacaftor, tezacaftor/ivacaftor/VX-659, tezacaftor/ivacaftor/VX-445 and tezacaftor/ivacaftor/VX-152) in clinical trials for patient with cystic fibrosis, according to age and mutation eligibility criteria.

Since 2016, the French patients homozygous for the p.Phe508del mutation and older than 12 years are able to be treated with the association LUMACAFTOR-IVACAFTOR and this French authorization is being extended for 6-11 years old children (while the European Commission has already granted an extension of the Marketing Authorization for lumacaftor/ivacaftor to include 6-11 years old children with cystic fibrosis since January 2018). Patients treated by lumacaftor/ivacaftor (or other ivacaftor new combinations) are closely monitored according to criteria established by the working group "New Therapeutic Approaches" of the French Society Cystic fibrosis.

This study is a phase IV observational trial for a period of 1 year. In this context, the team aims at initiating a comprehensive monitoring of the lung and gut mycobiota and microbiota evolution under LUMACAFTOR-IVACAFTOR (or other ivacaftor combinations) treatment. This project is directly linked to the monitoring of cystic fibrosis patients who begin treatment with LUMACAFTOR-IVACAFTOR (or other ivacaftor combinations) in France. The pro- and eukaryotic microbiota analysis is based on the secondary use of sputum and stool samples associated with several clinical data of CF patients under ivacaftor combinations and follow-up during the 1st year of therapy. According to the French law, Lum-Iva-Biota project is a non-interventional study. It aims at demonstrating that changes in the hydration of secretions at the pulmonary and intestinal levels related to LUMACAFTOR-IVACAFTOR therapy (or other new generation of ivacaftor combinations) promote a change in the lung and gut mycobiota and microbiota profiles which may achieve the characteristics of the "healthy type" (in terms of composition, richness and diversity).

DETAILED DESCRIPTION:
Cystic Fibrosis (CF) is related to structural and/or functional defects of chloride channel CFTR (Cystic Fibrosis Transport Regulator). These anomalies are associated with different classes of genetic mutations (class I to VI). The most common mutation is p.Phe508del class II (40% of homozygous and 70% heterozygous patients), it is responsible for the phenylalanine deletion at position 508 with improper intracellular processing of CFTR with less than normal amounts of CFTR protein at the apical cell membrane.

Over the last 20 years the CF patient outcome has been mainly improved using symptomatic treatments. More recently, new therapeutic strategies targeting directly CFTR defects have been developed. Initially potentiators which correct functional defects of CFTR (class Mutations 3 and 4) were studied. Then, correctors that target CFTR production were also developed. These molecules demonstrated substantial effect.

In 2015, the American company VERTEX - producing already KALYDECO (IVACAFTOR, VX-770) potentiator molecule that is recommended for the treatment of CF patients aged ≥ 6 y, with mutation altering the channel regulation (class III mutations) as G551D, G1244E, G1349D, G178R, G551S, S1251N, S1255P, S549Nou S549R) - was allowed by the Federal Drug Administration (FDA) and European Medicines Agency (EMA) for producing and using LUMACAFTOR-IVACAFTOR in clinical trials to manage CF patients over 12 years and having two p.Phe508del mutations. ORKAMBI represents the combination of two molecules (LUMACAFTOR + IVACAFTOR) respectively correctors and potentiator of CFTR.

This EMA authorization follows the results of two international studies (TRAFFIC and TRANSPORT) based on more than 1,000 CF patients showing that patients under LUMACAFTOR-IVACAFTOR compared to the group taking placebo have:

1. A moderate improvement in lung function (FEV1) at 24 weeks of 4.3 to 6.7%,
2. A significant reduction in lung exacerbations (bronchitis) up - 39%,
3. An increase in body mass index (BMI). These results confirm that LUMACAFTOR-IVACAFTOR may represent the first medicine to treat the whole underlying cause of CF in people ages 12 and older who have two copies of the p.Phe508del mutation. They complete the decrease or disappearance of pulmonary colonization with Pseudomonas aeruginosa (including mucoid phenotype isolates) observed under IVACAFTOR alone (KALYDECO treatment), even if the impact on fungal flora (or mycobiota) has not been described up to date.

In 2016, the French patients homozygous for the p.Phe508del mutation and older than 12 years were treated with this molecule association. Since January 2018, the European Commission has granted an extension of the Marketing Authorization for lumacaftor/ivacaftor to include 6 to 11 years old children with cystic fibrosis, and this authorization's extension is in process in France.

Since 2018 in France, VERTEX company has been allowed for producing and using new generations of ivacaftor combinations (tezacaftor/ivacaftor, tezacaftor/ivacaftor/VX-659, tezacaftor/ivacaftor/VX-445 and tezacaftor/ivacaftor/VX-152) in clinical trials for patient with cystic fibrosis, according to age (from 6 years old) and mutation eligibility criteria.

Patients treated by lumacaftor/ivacaftor or other ivacaftor combinations are closely monitored according to criteria established by the working group "New Therapeutic Approaches" of the French Society Cystic fibrosis. This study was a phase IV observational trial for a period of 1 year. In this context, the team aims at initiating a comprehensive monitoring of the lung and gut mycobiota and microbiota evolution under ivacaftor combinations (lumacaftor/ivacaftor or other ivacaftor combination).

This project is directly linked to the monitoring of homozygous p.Phe508del patients who begin treatment with ivacaftor combination in France (in agreement with the working group "New Therapeutic Approaches" of the French Society Cystic Fibrosis for lumacaftor/ivacaftor therapy, and the working group "Fungal Risks in CF").

As LUMACAFTOR-IVACAFTOR (or other ivacaftor combinations) impacts chloride secretion through CFTR at the apical site epithelial cells, with an expected improvement in secretion hydration and mucociliary clearance, it should modify the whole pulmonary microbial flora, including fungal microbiota (mycobiota) of CF lungs; this newly modified flora being expected achieving the characteristics of the "healthy type" in terms of flora composition, richness and diversity. We can expect same processes at the gut levels.

ELIGIBILITY:
Inclusion Criteria:

* CF Patient's ability to expectorate at inclusion time
* CF patient treated with an ivacaftor combination (lumacaftor/ivacaftor or new generation combination) for a period of at least 1 year and managed by the National working group "New therapeutic approaches" under the National CF Observatory and who haven't expressed a non-opposition to the secondary use of their sputum and stool samples in the context on Lum-Iva-biota project.

Exclusion Criteria:

* CF patient who stop ivacaftor combination treatment.
* CF patient who doesn't want to participate anymore to Lum-Iva-Biota

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: French patients with cystic fibrosis who start a treatment with an ivacaftor combination (lumacaftor/ivacaftor or new other combination) according to the age and mutations criteria in effect in France and monitored according to criteria established by the working group "New Therapeutic Approaches" of the French Society Cystic fibrosis.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Change of specific bacterial and/or fungal pathogens | 18 months
  Measure by conventional methods (history of microbial culture and GM assay) and particularly by metagenomic analysis of pulmonary pro- and eukaryotic microbiota.

SECONDARY OUTCOMES:
Forced expiratory volume in 1 second (FEV1) | Day 1
  Difference between the amount of air exhaled may be measured during the first second
Forced expiratory volume (FEV1) | 6 Months
  Difference between the amount of air exhaled may be measured during the first second
Forced expiratory volume (FEV1) | 12 Months
  Difference between the amount of air exhaled may be measured during the first second
Change of specific bacterial and/or fungal pathogens | 12 months
  Measure by conventional methods (history of microbial culture and GM assay) and particularly by metagenomic analysis of lung pro- and eukaryotic microbiota.
Change of specific bacterial and/or fungal pathogens | 12 months
  Measure by metagenomic analysis of gut pro- and eukaryotic microbiota.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence DELHAES, MD,PhD, Principal Investigator — University Hospital, Bordeaux
Locations (8):
- France (8):
  - CHU de Bordeaux - CRCM, Bordeaux
  - Centre Hospitalier Universitaire Grenoble Alpes, Grenoble
  - CHRU de Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - Assistance publique Hôpitaux Marseille, Marseille
  - Assistance Publique Hôpitaux de paris, Paris
  - Hôpital FOCH, Suresnes
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Enaud R, Lussac-Sorton F, Charpentier E, Velo-Suarez L, Guiraud J, Bui S, Fayon M, Schaeverbeke T, Nikolski M; LumIvaBiota Study Group; Burgel PR, Hery-Arnaud G, Delhaes L. Effects of Lumacaftor-Ivacaftor on Airway Microbiota-Mycobiota and Inflammation in Patients with Cystic Fibrosis Appear To Be Linked to Pseudomonas aeruginosa Chronic Colonization. Microbiol Spectr. 2023 Mar 27;11(2):e0225122. doi: 10.1128/spectrum.02251-22. Online ahead of print. PMID 36971560